CLINICAL TRIAL: NCT00191269
Title: A Multicenter Study of LY188011 in Anthracyclines and Taxanes Pre-treated Metastatic/Recurrent Breast Cancer
Brief Title: Gemcitabine Monotherapy for Metastatic Breast Cancer After Anthracycline and Taxane Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9065; B9E-JE-MB21 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-05-14 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Metastatic Breast Cancer
Keywords: after; anthracycline; taxane; regimen
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Dose Level 1 - 1000 mg/m2
  Interventions: Drug: gemcitabine
- B (Experimental): Dose Level 2 - 1250 mg/m2
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — 1000 mg/m2, intravenous (IV), day 1 and day 8 every 21 days
  Other Names: LY188011; Gemzar
  Arms: A
Drug: gemcitabine — 1250 mg/m2, intravenous (IV), day 1 and day 8 every 21 days
  Other Names: LY188011; Gemzar
  Arms: B

SUMMARY:
To investigate efficacy, safety and PK of GEM monotherapy after prior chemotherapy with anthracycline and taxane regimen for patients with metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed breast cancer
* Received prior chemotherapy for metastatic breast cancer with anthracycline and taxane regimen
* To have at least one measurable region
* PS: 0-1
* To have adequate organ function (bone marrow, liver and renal function)

Exclusion Criteria:

* To have Interstitial pneumonia or pulmonary fibrosis
* To have inflammatory carcinoma
* Within 28 days after the latest chemotherapy or radiotherapy, 14 days after the latest hormonal/immunotherapy or 7 days after surgery
* To have brain metastasis with symptom
* To have severe complication (cardiac infarction, infection, drug hyper sensitivity or diabetes)

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Japan (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Step 1, 6 participants each were assigned at Dose Level 1 (gemcitabine:1000 mg/ m2) and Dose Level 2 (gemcitabine:1250 mg/ m2) to determine the recommended dose for Step 2. At Step 2, an additional 56 participants received the recommended dose (Dose Level 2).
Groups:
- Dose Level 1: Gemcitabine at 1000 mg/m2 administered intravenously over 30 to 60 minutes on Days 1 and 8 in each 3-week (21-day) cycle of study therapy.
- Dose Level 2: Gemcitabine at 1250 mg/m2 administered intravenously over 30 to 60 minutes on Days 1 and 8 in each 3-week (21-day) cycle of study therapy.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 6 | 62
Completed | 0 | 4
Not Completed | 6 | 58
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 1 | 4
Not completed — Progression of Disease | 4 | 42
Not completed — Lack of Efficacy | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Pathologic Aggrevation | 0 | 1
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 6 | 62 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 53.3 (7.45) | 52.4 (11.25) | 52.5 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 62 | 68.0
  Male | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 62 | 68.0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 4 | 45 | 49.0
    1 - Ambulatory, Restricted Strenuous Activity | 2 | 17 | 19.0
Human Epidermal Growth Factor Receptor 2 Expression Status [Number; unit: participants]
  0 | 2 | 27 | 29.0
  1+ | 1 | 20 | 21.0
  2+ | 2 | 4 | 6.0
  3+ | 1 | 9 | 10.0
  Unknown | 0 | 2 | 2.0
Presence of Estrogen Hormone Receptor [Number; unit: participants]
  None | 4 | 25 | 29.0
  Present | 2 | 37 | 39.0
  Unknown | 0 | 0 | 0.0
Presence of Metastasis [Number; unit: participants] — Metastasis could occur in more than one site, resulting in a higher sum for all categories in the arm/group than the overall number of participants in the arm/group.
  participants
    None | 0 | 5 | 5.0
    Lung | 0 | 27 | 27.0
    Bone | 1 | 24 | 25.0
    Liver | 2 | 25 | 27.0
    Brain | 0 | 0 | 0.0
    Lymph Node | 2 | 23 | 25.0
    Skin | 1 | 6 | 7.0
    Other Sites | 0 | 13 | 13.0
Presence of Progesterone Hormone Receptor [Number; unit: participant]
  None | 3 | 39 | 42.0
  Present | 2 | 23 | 25.0
  Unknown | 1 | 0 | 1.0
Time of Latest Chemotherapy Completion [Number; unit: participants]
  <3 months | 2 | 40 | 42.0
  ≥3 months and <6 months | 1 | 6 | 7.0
  ≥6 months and <1 year | 3 | 9 | 12.0
  ≥1 year and <2 years | 0 | 3 | 3.0
  ≥2 years and <3 years | 0 | 2 | 2.0
  ≥3 years before | 0 | 2 | 2.0
Time to Recurrence [Number; unit: participants]
  <1 year | 4 | 22 | 26.0
  ≥1 year and <2 years | 0 | 18 | 18.0
  ≥2 years and <3 years | 0 | 4 | 4.0
  ≥3 years and <4 years | 0 | 2 | 2.0
  ≥4 years and < 5 years | 0 | 2 | 2.0
  ≥5 to <10 years | 1 | 4 | 5.0
  No Recurrence | 1 | 10 | 11.0
Height [Mean (Standard Deviation); unit: centimeters] | 152.45 (4.05) | 156.43 (6.04) | 156.08 (5.98)
Weight [Mean (Standard Deviation); unit: kilograms] | 47.73 (1.46) | 57.02 (9.15) | 56.20 (9.13)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: baseline to measured progressive disease
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 62
participants
  Complete Response | 0 | 1
  Partial Response | 0 | 4
  Long Stable Disease | 1 | 4
  Stable Disease | 1 | 16
  Progressive Disease | 2 | 32
  Not Evaluable | 2 | 5

2. Secondary Outcome: Duration of Response
Description: For responders, the minimum and maximum of the duration of complete response, duration of partial response, and duration of overall response were summarized, and the median of response duration and its 95% confidence interval were calculated using the Kaplan-Meier estimation.
Time Frame: time of response to progressive disease
Population: The 5 responding participants (complete response and partial response) at Dose Level 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 5
months |  | 10.07 [5.43 to 13.80]

3. Secondary Outcome: Time to Progressive Disease
Description: Time from study enrollment to first date of disease progression. Time to disease progression was censored at date of death if death was due to other cause. The minimum and maximum of this parameter were summarized, and the median time to progression and its 95% confidence interval were calculated using the Kaplan-Meier estimation.
Time Frame: baseline to measured progressive disease
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 62
days | 137 [97 to 196] | 92 [78 to 121]

4. Secondary Outcome: Survival at 1 Year
Description: Results are reported as number of participants alive at one year.
Time Frame: baseline to date of death from any cause, evaluate at 1 year
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 62
participants | 4 | 42

5. Secondary Outcome: Pharmacokinetics - Normalized Cmax
Description: maximum gemcitabine plasma concentration normalized to 1250 milligrams per square meter of gemcitabine.
Time Frame: cycle 1
Population: Pharmacokinetic data were available from 12 patients.
Measure: Geometric Mean (Full Range); unit: nanograms per milliliter (ng/mL)
Groups:
- Dose Normalized to 1250 Milligrams Per Square Meter: 12 participants with a mean gemcitabine dose of 1120 milligrams per square meter
Arm/Group | Dose Normalized to 1250 Milligrams Per Square Meter
Number analyzed (Participants) | 12
nanograms per milliliter (ng/mL) | 29,036 [16,341 to 53,857]

6. Secondary Outcome: Pharmacokinetics - Normalized Area Under the Curve
Description: Area under the gemcitabine plasma concentration-time curve from time zero to infinity. Gemcitabine dose was normalized to 1250 milligrams per square meter.
Time Frame: cycle 1
Population: Pharmacokinetic data were available on 12 participants.
Measure: Geometric Mean (Full Range); unit: nanograms times hour per milliliter
Arm/Group | Dose Normalized to 1250 Milligrams Per Square Meter
Number analyzed (Participants) | 12
nanograms times hour per milliliter | 15,999 [9,929 to 21,723]

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 1 | 10
Other Adverse Events (participants affected / at risk) | 4 | 34
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Dose Level 1 | Dose Level 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 0/62 (0)
Cellulitis (Infections and infestations) | 1/6 (1) | 1/62 (1)
Blood lactate dehydrogenase increased (Investigations) | 0/6 (0) | 1/62 (1)
Catheterisation venous (Surgical and medical procedures) | 0/6 (0) | 2/62 (2)
Infection (Infections and infestations) | 0/6 (0) | 1/62 (1)
Femur fracture (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/62 (1)
Cardiac failure acute (Cardiac disorders) | 0/6 (0) | 1/62 (1)
Anorexia (Metabolism and nutrition disorders) | 0/6 (0) | 1/62 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/62 (1)
Brain oedema (Nervous system disorders) | 0/6 (0) | 1/62 (1)
Cataract (Eye disorders) | 0/6 (0) | 1/62 (1)
Raynaud's phenomenon (Vascular disorders) | 0/6 (0) | 1/62 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Dose Level 1 | Dose Level 2
Alanine aminotransferase increased (Investigations) | 1/6 (1) | 8/62 (8)
Neutrophil count decreased (Investigations) | 2/6 (2) | 26/62 (26)
Anorexia (Metabolism and nutrition disorders) | 1/6 (1) | 1/62 (1)
Nausea (Gastrointestinal disorders) | 0/6 (0) | 3/62 (3)
Vomiting (Gastrointestinal disorders) | 0/6 (0) | 3/62 (3)
Malaise (General disorders) | 0/6 (0) | 1/62 (1)
Pyrexia (General disorders) | 0/6 (0) | 1/62 (1)
Nasopharyngitis (Infections and infestations) | 0/6 (0) | 1/62 (1)
Aspartate aminotransferase increased (Investigations) | 0/6 (0) | 4/62 (4)
C-reactive protein increased (Investigations) | 0/6 (0) | 1/62 (1)
White blood cell count increased (Investigations) | 0/6 (0) | 1/62 (1)
Dizziness (Nervous system disorders) | 0/6 (0) | 1/62 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/62 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/62 (1)
Tooth extraction (Surgical and medical procedures) | 0/6 (0) | 1/62 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days